CLINICAL TRIAL: NCT05611528
Title: Safety and Effectiveness of Evinacumab for the Treatment of Homozygous Familial Hypercholesterolemia in a Real Life Setting in Canada
Brief Title: Safety and Effectiveness of Evinacumab for the Treatment of Homozygous Familial Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daniel Gaudet (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor-Investigator, Daniel Gaudet, Director, Ecogene 21
Organization: Ecogene 21 (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECO HoFH-2022-01
Record Dates: First submitted 2022-10-31; First posted 2022-11-10 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Homozygous Familial Hypercholesterolemia
Keywords: ANGPTL3; Real-life study; Monoclonal antibody
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — evinacumab

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Evinacumab-treated patients (Experimental)
  Interventions: Drug: Evinacumab

INTERVENTIONS:
Drug: Evinacumab — Evinacumab 15 mg/kg administered intravenously every 4 weeks

SUMMARY:
This is an open-label study designed to evaluate the long-term safety and efficacy of evinacumab, a fully human ANGPTL3 antibody, in patients with homozygous familial hypercholesterolemia (HoFH), in a real-life setting in Canada.

Eligible patients for this study are male and female adult patients with HoFH. Evinacumab will be added on top of the patient's background lipid-modifying therapy (LMT), including statins, ezetimibe, PCSK9 inhibitors, lomitapide or other lipid lowering therapies. This study will be conducted using an hybrid (on-site, foldable sites) approach. Patients will enter the current study, in an open-label treatment period, following their screening. This study will continue until reimbursement of evinacumab in Canada or for a maximum of 24 months. The end of study (EoS) visit will be scheduled 4 weeks after the last dose has been injected and will be followed by a 52-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* HoFH patients having been previously or being currently treated with evinacumab or clinical diagnosis of HoFH requiring additional lipid lowering therapy.

Exclusion Criteria:

* Any new condition or worsening of an existing condition, which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study;
* Pregnant or breastfeeding women;
* Women of childbearing potential who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 24 weeks after the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Change in lipid profile | Every 4 weeks up to 2 years
  Change in total cholesterol, LDL-Cholesterol, HDL-Cholesterol, triglyceride, non-HDL-Cholesterol and apolipoprotein B plasma concentration
Change in aspartate transaminase (AST) plasma concentration | Every 4 weeks up to 2 years
change in alanine aminotransferase (ALT) plasma concentration | Every 4 weeks up to 2 years

SECONDARY OUTCOMES:
Lipoprotein (a) | Yearly up to 2 years
Complete blood count | Every 12 weeks up to 2 years
Total bilirubin | Every 12 weeks up to 2 years
Creatine phosphokinase | Every 12 weeks up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ecogene-21, Saguenay, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided